CLINICAL TRIAL: NCT04804488
Title: Recurrent Nasal Polyposis; A Two Years Retrospective Comprehensive Overview
Brief Title: Retrospective Study for Recurrent Nasal Polyposis
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shimaa Rafaat Mohamed, M.B.B.Ch, resident of Otorhinolaryngology at Sohag General Hospital, Sohag University
Other Study IDs: Soh-Med-21-01-03
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Nasal Polyps
MeSH Terms: conditions — Nasal Polyps

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: nasal polyp surgery — A retrospective study for patients with recurrent nasal polypi operated at Otorhinolaryngology Department, Sohag University Hospital will be carried out.

SUMMARY:
A retrospective study for patients with recurrent nasal polypi operated at Otorhinolaryngology Department, Sohag University Hospital will be carried out.

DETAILED DESCRIPTION:
A retrospective study for patients with recurrent nasal polypi operated at Otorhinolaryngology Department, Sohag University Hospital will be carried out. All available information about these patients will be retrieved from our department data base including full personal history, medical history and type of surgery performed with operative details.. Missed patients due to any reason will be excluded from the study during. Complete information about patients' symptoms, onset, progression, severity and duration of recurrence after surgery will be taken from our department data base. Associated factors will be evaluated from data base (asthma, allergy, smoking, Samter's triad, cystic fibrosis, fungal sinusitis, immune status, etc.).

ELIGIBILITY:
Inclusion Criteria:

All patients with recurrent nasal polypi will be include in our study regardless their age and sex.

Exclusion Criteria:

* Exclusion criteria:

Patients with nasal polyps due to underlying neoplasm will be excluded from our study. Also, those with fresh polyps or missed patients during follow up due to any reason are not candidates for our research.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: To evaluate patients with recurrent nasal polypi operated at Otorhinolaryngology department, Sohag University Hospital during the period from July 2018 to July 2020, discuss their epidemiologic aspects, management and outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Recurrent Nasal Polyposis | A Two Years Retrospective Comprehensive Overview
  Aim of the work:
  To evaluate patients with recurrent nasal polypi operated at Otorhinolaryngology department at sohag university hospital

CONTACTS AND LOCATIONS:
Overall Officials: shimaa R Mohamed, master, Principal Investigator — M.B.B.Ch, resident of Otorhinolaryngology at Sohag General Hospital
Locations (1):
- Sohag University hospital, Sohag, Egypt